CLINICAL TRIAL: NCT02703948
Title: Injection Technique Assessment of Restylane Silk With Lidocaine for Lip Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43USC1505
Record Dates: First submitted 2016-03-03; First posted 2016-03-09 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2018-04

CONDITIONS: Lip Augmentation and Correction of Perioral Rhytids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restylane Silk with Lidocaine (Other)
  Interventions: Device: Restylane Silk with Lidocaine

INTERVENTIONS:
Device: Restylane Silk with Lidocaine

SUMMARY:
This is a multi-center, open-label, single-arm study to assess the safety of an injection technique with Restylane Silk in lip augmentation and correction of perioral rhytids .

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to comply with the requirements of the study and providing written informed consent including release of copyright of photography images.
* Males or females, 22 years of age or older
* Subjects seeking augmentation therapy for the lips.

Exclusion Criteria:

* History of allergy or hypersensitivity to injectable HA gel or to gram positive bacterial proteins.
* History of allergy or hypersensitivity to lidocaine, other amide type anesthetics, or topical anesthetics or nerve blocking agents
* Previous surgery to the upper or lower lip, lip piercing or tattoo, or history of facial trauma.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - United States, California, Beverly Hills, California
  - United States, California, San Diego, California
  - United States, Florida, Miami, Florida
  - United States, Georgia, Roswell, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Restylane Silk With Lidocaine: Restylane Silk with Lidocaine
Period: Overall Study
Arm/Group | Restylane Silk With Lidocaine
Started | 60
Completed | 57
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Restylane Silk With Lidocaine
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 53
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events With the Use of Restylane Silk With Lidocaine
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Silk With Lidocaine
Number analyzed (Participants) | 60
Participants | 11

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from screening through 12 weeks
Arm/Group | Restylane Silk With Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 11/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Silk With Lidocaine (N=60)
Bruising (General disorders) | 4 (5)
Pain (General disorders) | 1 (2)
Swelling (General disorders) | 8 (14)
Chapped Lips (Gastrointestinal disorders) | 1 (2)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any and all data resulting from the Study will not be presented or published in any form or media by the PI without the prior written consent of the Sponsor.